CLINICAL TRIAL: NCT03111706
Title: 2D and 3D Ultrasound Assessment of Cesarean Section Scars and Its Correlation to Intraoperative Findings
Brief Title: 2D and 3D Ultrasound Assessment of Cesarean Section Scars
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Other Study IDs: 165
Record Dates: First submitted 2017-04-08; First posted 2017-04-13 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Cesarean Wound Disruption
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dehiscencd scar: women who are discovered with scar dehiscence during cesarean section
  Interventions: Procedure: Cesarean section
- Intact scar: women with intact scar detected during cesarean section
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Procedure: Cesarean section — During Cesarean delivery the lower uterine segment (LUS) was defined as the part of the uterus below the uterovesical peritoneal reflection. After opening the visceral peritoneum and performing the bladder dissection, the LUS was assessed for integrity of the CS scar by the operating surgeon to avoid bias by the sonographic findings. Scar dehiscence was defined as the presence of either transparent LUS with visible contents, presence of well-circumscribed scar defect or presence of frank uterine rupture.

SUMMARY:
Prospective observational study conducted on women with previous 1 or 2 CS candidate for elective CS. Ultrasonographic evaluation of lower uterine segment using 2D and 3D transabdominal and transvaginal then correlated to scar integrity assessed intraoperatively

DETAILED DESCRIPTION:
Transabdominal ultrasound examination to obtain full obstetric ultrasound report including estimated gestational age, fetal lie, presentation, amniotic fluid volume, placental location with special focus on relation to the uterine scar.

The second step was to measure the thickness of the LUS using 2D ultrasound. View of the LUS was obtained in the mid-sagittal plane and the view was magnified looking for the thinnest area of the LUS. Also, the LUS was examined in a lateral view to detect any apparent rupture, ballooning or funneling. The measurement was taken with the cursors at the urine-Urinary bladder interface and the amniotic fluid -decidua interface after sufficient magnification and measurement was taken to the nearest tenth of millimeter. The numeric display was covered during the examination to avoid bias when performing the 3D measurement in the next step. Three measurements were taken and the least measurement was recorded.

After the entire thickness was measured by 2D ultrasound, 3 D measurement were taken in the mid-saggittal plan using the multiplanar display mode and then moving through the acquired 3-D volume in the saggittal plane till the thinnest area was seen and then measurements were taken.3-D volume dataset was obtained of the LUS by the same operator. The acquired volume was manipulated on the multiplanar display mode, searching for the thinnest part of the LUS avoiding obliquity.

Transvaginal ultrasound examination was done following the transabdominal one. The vaginal probe was inserted into the posterior vaginal fornix with the patient lying supine and the patient's knees are gently flexed and hips are slightly elevated with a pillow. Clear view of the LUS was obtained in the midsagittal plane visualizing the cervical canal to ensure that the view is midline one and avoiding obliquity.

On transvaginal examination the muscular layer of the LUS was clearly seen as hypoechoic line between the hyperechoic uterovesical fold and the decidualized endometrium and the chorioamniotic membranes. The scar area was magnified so the scar occupies at least 75% of the image to ensure consistent and accurate measurements. The thickness of the muscular layer of LUS was taken with the measuring caliber placed at the urinary bladder wall-myometrium interface and the myometrial/ chorioamniotic membrane interface .Three measurements of the LUS were taken, and again, the least measurement was recorded.

Again, 3D volume data set of the LUS was obtained .The acquired volume was manipulated on the multiplanar display looking for the thinnest part of the muscular layer. The thickness was measured to the nearest tenth of millimeter and recorded. The same operator has performed the transabdominal and transvaginal sonographic examination, and the surgeon performing the CS was always blinded of the sonographic findings.

The ultrasound examination to CS time interval varied from one to forty eight hours. During Cesarean delivery the LUS was defined as the part of the uterus below the uterovesical peritoneal reflection. After opening the visceral peritoneum and performing the bladder dissection, the LUS was assessed for integrity of the CS scar by the operating surgeon to avoid bias by the sonographic findings. Scar dehiscence was defined as the presence of either transparent LUS with visible contents, presence of well-circumscribed scar defect or presence of frank uterine rupture.

ELIGIBILITY:
Inclusion Criteria:

* 37 - 40 weeks of gestational age
* singleton pregnancy,
* cephalic presentation,
* not in labor
* intact membranes
* with history of one or two previous CS

Exclusion Criteria:

* disorders of amniotic fluid,
* placenta previa
* history of other uterine surgery, e.g, myomectomy

Ages: 19 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: women with prior 1 or 2 cesarean sections candidate for elective cesarean sewction
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Scar dehiscence | At time of surgery
  as the presence of either transparent LUS with visible contents, presence of well-circumscribed scar defect or presence of frank uterine rupture.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided